CLINICAL TRIAL: NCT04402528
Title: Improving Rates of Behavioral Treatment in Preschoolers Through Mehealth for ADHD Software
Brief Title: Preschool ADHD On-line Behavioral Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Developmental Behavioral Pediatrics Research Network (Unknown); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Tanya Froehlich, MD, Professor of Pediatrics and Director of Research, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1274
Record Dates: First submitted 2020-04-24; First posted 2020-05-27 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mehealth portal with integrated behavioral tools (Experimental): Patients in this arm will use the mehealth for ADHD web-based software and have access to a module that allows parents and teachers/childcare providers to develop and implement behavioral interventions such as daily report cards online.
  Interventions: Behavioral: Behavioral tools integrated within mehealth for ADHD software

INTERVENTIONS:
Behavioral: Behavioral tools integrated within mehealth for ADHD software — Integrated functionality within the mehealth for ADHD software allows parents and teachers/childcare providers to set up and deliver behavioral interventions such as daily report card systems and home-based program such as star charts. Automated wizards lead parents and teachers through the process of selecting target behaviors and setting up reward schedules. Baseline data is gathered online and algorithms derive a set of behavioral goals for the child. Thereafter, parents or teachers record the child's performance directly into the software. Once behavioral monitoring begins, parents and teachers receive daily email or text communications from mehealth for ADHD alerting them to the daily rewards earned by their child. Finally, online algorithms exist that detect how a child is doing in meeting behavioral goals and prompt users to modify goals accordingly.
  Other Names: mehealth for ADHD

SUMMARY:
The primary goal of the proposed project is to test the feasibility of parent and teacher/childcare providers use of the ADHD web portal-integrated behavioral treatment modules with preschool children with ADHD in order to improve the access to and the integrity of evidence-based behavioral treatment strategies for young children with ADHD.

DETAILED DESCRIPTION:
Although behavioral interventions are the recommended first-line treatment for preschool children with Attention Deficit Hyperactivity Disorder (ADHD), the majority of preschool children receiving treatment for ADHD are treated with medication only. Barriers to preschool children receiving behavioral treatments include financial limitations, family logistical challenges, and the paucity of trained providers. Web-based approaches may be one innovative way to address these obstacles. Thus, the goal of the proposed study is to pilot-test an on-line behavioral intervention that has been integrated into the evidence-based mehealth for ADHD software (mehealth.com) to determine feasibility, acceptability, and preliminary efficacy. The investigators will enroll a community-based sample of caregivers and teachers/childcare providers of 20 preschool children with ADHD recruited from two DBPNet sites (Cincinnati and Boston) who will utilize the on-line behavioral tools to create and implement child behavior plans. The investigators will track system usage over a 9-month period to determine feasibility for mehealth's integrated behavioral tools intervention. Standardized measures and open-ended questions will be used to determine the intervention's acceptability to parents and teachers/childcare providers. In addition, parent and teacher/childcare providers ratings of child ADHD symptoms and impairment collected at baseline and at the 3-month, 6-month, and 9-month time points will be examined to provide preliminary estimates of efficacy. Ultimately, development of the mehealth for ADHD.com integrated behavioral tools may provide a cost-effective and convenient means of implementing behavioral plans for young children, thereby increasing access to behavioral treatments for preschoolers with ADHD. This scalable and disseminatable approach has great potential for use not only in clinical settings, but also in national Developmental-Behavioral Pediatrics Research Network multi-site research studies which require standardized behavioral intervention packages for preschool ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Child has been diagnosed with ADHD, or shows significant signs and symptoms of ADHD.
* If child is being prescribed ADHD medication, child must currently be on a stable dosage of medication for 1 month.
* Child meets criteria for a research diagnosis of ADHD* based on the ADHD Rating Scale IV Preschool-Version and Impairment Rating Scale assessments that the parent completes.

  * Children will be given a research diagnosis of ADHD if the following criteria are met: 1) parents endorse that children have 6 or more symptoms in either the inattentive or hyperactive-impulsive domains present "often" or "very often" on the ADHD Rating Scale IV-Preschool Version (ADHD-RS-IV-P) or Vanderbilt ADHD Rating Scale; or have inattentive symptom scores and/or hyperactive symptom scores >93th percentile for sex on the ADHD-RS-IV-P AND 2) child is experiencing ADHD-related impairment as shown by the parent or a teacher/childcare provider/additional adult scoring one or more items on the Impairment Rating Scale as a 3 or higher. Note: child behavior ratings from a teacher/childcare provider/additional adult on the ADHD-RS-IV-P and Impairment Rating Scale will not be required for study inclusion and children will not be excluded from the study on the basis of these ratings. Parents of children with a research diagnosis of ADHD will be eligible for study participation.

Exclusion Criteria:

* Parent does not have access to a computer or smartphone.
* Child has global developmental delay.
* Child has been diagnosed with autism spectrum disorder.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
% of days using mehealth behavior tracking system | 9 months
  Feasibility will be assessed by tracking system usage, including % of days when parents/teachers/childcare providers entered behavioral tracking data (to determine if data was entered for >85% of days) and % of days when earned rewards were administered (to determine if administration occurred for >85% of days).
Acceptability with on-line behavioral treatment assessed by the System Usability Scale | 9 months
  System Usability Scale contains ten items rated on a Likert scale.
  - SUS contains ten items rated on a Likert scale.
  Acceptability with on-line behavioral treatment assessed by the Intervention Acceptability Questionnaire (IAQ).
  - The IAQ contains 3 open-ended questions regarding satisfaction with the on-line behavioral treatment program.
Acceptability with on-line behavioral treatment assessed by the Intervention Acceptability Questionnaire | 9 months
  The Intervention Acceptability Questionnaire contains 3 open-ended questions regarding satisfaction with the on-line behavioral treatment program

SECONDARY OUTCOMES:
ADHD Rating Scale-IV-Preschool Version | 9 months
  Descriptive statistics from parent-rated ADHD Rating Scale-IV-Preschool Version total symptom scores will be reported across time points. Please note that the word "ADHD" is not used as an abbreviation in "ADHD Rating Scale - IV - Preschool Version," that is the official name of the scale.
Impairment Rating Scale | 9 months
  Descriptive statistics from parent-rated Impairment Rating Scale total symptom scores will be reported across time points

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Froehlich, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No